CLINICAL TRIAL: NCT01885663
Title: Umbilical Cord Blood Therapy for Patients With Acquired Brain Injury
Brief Title: UCB Therapy in Acquired Brain Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MinYoung Kim, M.D. (Other)
Responsible Party: Sponsor-Investigator, MinYoung Kim, M.D., Professor, Bundang CHA Hospital
Organization: Bundang CHA Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCBABI
Record Dates: First submitted 2013-06-20; First posted 2013-06-25 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Acquired Brain Injury
Keywords: Umbilical cord blood; Acquired brain injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: UCB therapy for TBI patient
Oversight: Data Monitoring Committee: No

ARMS (1):
- Umbilical cord blood therapy (Experimental): Umbilical cord blood therapy
  Interventions: Procedure: Umbilical cord blood therapy

INTERVENTIONS:
Procedure: Umbilical cord blood therapy — Intravascular umbilical cord blood therapy

SUMMARY:
This open label trial is conducted to investigate the efficacy and safety of allogeneic umbilical cord blood (UCB) therapy for patients with acquired brain injury.

DETAILED DESCRIPTION:
Acquired brain injury (ABI) means brain damage caused by events after birth, rather than as part of a genetic or congenital disorders. Those with ABI suffer from cognitive, physical, or behavioral impairments limiting their activity and participation in society. ABI results from traumatic or non-traumatic brain injury due to internal or external source (e.g. infection, brain tumor, hypoxia). Preclinical studies regarding cell therapy in animal models of ABI showed improvements of neurological dysfunction. UCB possess various stem or progenitor cells and is known to secrete neurotrophic factors to repair injured brain. This clinical research aims to determine the safety and efficacy of allogeneic UCB for patients with ABI.

ELIGIBILITY:
Inclusion Criteria:

* Acquired brain injury
* Duration: over 12 months
* Willing to comply with all study procedure

Exclusion Criteria:

* Medical instability including pneumonia or renal function at enrollment
* Uncontrolled persistent epilepsy
* Poor cooperation of guardian,including inactive attitude for rehabilitation and visits for follow-up
* Not eligible according to the principal investigator

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2013-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Monitoring adverse events | 12 months

SECONDARY OUTCOMES:
Changes in standardized gross motor function | Baseline - 1 month - 3 months - 6 months - 12 months
  GMFM (Gross Motor Function Measure) as a standardized measurement tool for assessing Gross Motor Function consisting of sub-scales; lying & rolling, sitting, crawling & kneeling, standing, walking, running & jumping (range: 0~100 , Higher value means better gross motor function.)
Changes in motor performance | Baseline - 1 month - 3 months - 6 months - 12 months
  GMPM (Gross Motor Performance Measure) as a standardized measurement tool for assessing quality of movement regarding 3 properties of 5 ones; alignment, coordination, dissociated movement, stability, and weight shift (range: 0~100, Higher value means better motor quality.)
Changes in cognitive neurodevelopmental outcome | Baseline - 1 month - 3 months - 6 months - 12 months
  Korean version of Bayley Scale of Infant Development-II Mental Scales (Higher value means better cognitive function: raw score 0 - worst, 178 - best.)
Changes in motor neurodevelopmental outcome | Baseline - 1 month - 3 months - 6 months - 12 months
  Korean version of Bayley Scale of Infant Development-II Motor Scales (Higher value means better motor function: raw score 0 - worst, 112 - best)
Changes in functional performance in daily activities | Baseline - 1 month - 3 months - 6 months - 12 months
  Pediatric Evaluation of Disability Inventory (PEDI) for assessing functional performance in daily activities in children (All values are adjusted and higher value means better functional performance, 0 - worst, 100 - best.)
Changes in brain glucose metabolism | Baseline - 12 months
  FDG (fludeoxyglucose)-PET (positron emission tomography)
Changes in brain white matter integrity | Baseline - 12 months
  diffusion tensor imaging

CONTACTS AND LOCATIONS:
Overall Officials: MinYoung Kim, M.D., Ph.D., Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea